CLINICAL TRIAL: NCT03394066
Title: Understanding the Acute Modulation of Brain Activity by Transcranial Magnetic Stimulation
Brief Title: Mechanism of Non-invasive Magnetic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 999918042; 18-DA-N042
Record Dates: First submitted 2018-01-06; First posted 2018-01-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12-18

CONDITIONS: Healthy Volunteers
Keywords: Repetitive TMS (rTMS); Simultaneous TMS and MRI
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TMS (Experimental): All participants will receive TMS to investigate acute modulations of brain activity by TMS
  Interventions: Device: TMS (MagVenture MagPro 100 with MagOption)

INTERVENTIONS:
Device: TMS (MagVenture MagPro 100 with MagOption) — TMS will be applied using the MagVenture MagPro 100 with MagOption (MagVenture Inc, Alpharetta, GA) stimulator with a figure-of-eight TMS coil. An MRI compatible version of the figure-of-eight coil will be used inside the MRI scanner with an appropriate TMS coil holder.

SUMMARY:
Background:

Transcranial magnetic stimulation (TMS) is form of non-invasive brain stimulation. It is approved to treat depression. TMS may help decrease drug craving. It is important to understand how TMS affects the brain. Such a better understanding would help to design ways to treat drug addiction.

Objectives:

To learn how TMS affects the brain when it stimulates an area in the front of the brain. Also, to see how the stimulation affects the area stimulated and other connected areas.

Eligibility:

Healthy, right-handed adults ages 18-60 who are non-drug users.

Design:

Participants will be screened under protocol 06-DA-N415.

Participants will have at least 3 visits. The first visit will last about 3 hours. All other visits will last up to 6 hours. Participants cannot use drugs or alcohol at least 24 hours before a visit. They cannot have more than half a cup of a caffeinated drink at least 12 hours before a visit.

Each visit will include a brief medical history update, urine test for drugs and pregnancy (if female), a breath test for alcohol and smoking, and questionnaires.

Participants will have a TMS orientation visit. A wire coil will be placed on the head. An electrical current will pass through the coil to create a magnetic pulse that stimulates the brain.

The other visits will include 2 sessions of TMS-MRI. Participants will lie on a table that slides into a cylinder. The TMS coil and the MRI coil will be placed over the head. Pictures will be taken of the brain with and without stimulation.

Participants will complete a questionnaire about how they feel before and after each TMS session and in a follow-up call 2-3 weeks after their last session.

DETAILED DESCRIPTION:
Objectives:

The goal of the protocol is to investigate acute modulations of brain activity by transcranial magnetic stimulation (TMS). Using simultaneous TMS and functional magnetic resonance imaging (fMRI), we will evaluate TMS induced changes in brain activity, including regional brain activation and inter-regional functional connectivity. Repetitive TMS will be applied over the dorsolateral prefrontal cortex (DLPFC) with different frequencies and interleaved with fMRI acquisition to provide online monitoring of brain activity. Furthermore, we will assess the relationship between the TMS induced brain activity and the anatomical connection obtained from diffusion tensor imaging (DTI), using individual variations in these imaging measures. Results from this study will help to understand the underling mechanism of TMS and will provide insights for interpretation of TMS and fMRI data.

Study population:

Up to 70 healthy, adults will be tested. Subjects must fit exclusion/inclusion criteria for both TMS and MRI. We expect to enroll 70 subjects to arrive at 50 who complete the protocol.

Design:

The study is a within-subject design with each subject completing up to 6 TMS-fMRI sessions in three days (2 sessions per day)

Outcome measures:

The outcome measures will be the effects of TMS on fMRI blood oxygen level-dependent (BOLD) responses, TMS induced changes on resting state functional connectivity, and their associations with relevant structural connectivity revealed by DTI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must:

1. Be 18 - 60 years of age.

   -Justification: Many neural processes change with age, and these changes could introduce unwanted variability in both behavioral and MRI signals. In addition, the risk of difficult-to-detect medical abnormalities such as silent cerebral infarcts increases with age.

   --Screening tool: History.
2. Be in good health.

   * Justification: Many illnesses may alter neural functioning as well as fMRI signals.
   * Screening tools: Medical Assessment, Medical History and Physical Examination. Medical assessments include: Vital Signs, oral HIV test, height/weight measurements, and blood sample. Tests on the blood sample include CBC, Hemoglobin A1C, complete metabolic profile, ESR, and HIV (if needed to confirm a positive salivary test for HIV). The following individual laboratory results will independently disqualify individuals: Hemoglobin < 10.5 g/dl, Hemoglobin A1C >6.5%, WBC < 2400/microliter, LFTs > 3Xnormal, and Casual serum glucose > 200 mg/dl. The MAI will retain discretion to exclude at less extreme values, depending on the clinical presentation. Elevated serum glucose may be followed up to assess for diabetes. MAI will make the final judgment on any questionable lab results.
3. Right-handed.

   * Justification: Using right-handed individuals will reduce variability in BOLD MRI data.
   * Screening tool: self-report.

EXCLUSION CRITERIA:

1. Personal history of stroke, brain lesions, previous neurosurgery, any personal history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than two days.

   * Justification: Stroke or head trauma can lower the seizure threshold and are therefore contraindications for TMS. Fainting episodes or syncope of unknown cause could indicate an undiagnosed condition associated with seizures. Neurological symptoms could potentially alter BOLD signal.
   * Screening tool: TMS safety questionnaire and History and Physical including a neurological exam.
2. First-degree family history of any form of epilepsy with a potentially hereditary basis.

   * Justification: First-degree family history of epilepsy with a hereditary component increases the risk of the participant having an undiagnosed condition that is associated with lowered seizure threshold.
   * Screening tool: TMS safety screening, Medical History.
3. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, -shunts, stimulators, cochlear implants, or electrodes) or any other metal object in the body that precludes either MRI scanning or TMS intervention.

   * Justification: Any metal around the head is a contraindication for both MRI and TMS, as both methods involve exposure to a relatively strong magnetic field.
   * Screening tool: TMS safety screening, MRI safety screening, Medical History.
4. Any contraindications to MRI or TMS.

   * Justification: There are additional contraindications that would exclude participation in MRI or TMS (e.g., claustrophobia).
   * Screening tool: MRI safety screening, TMS Safety Screening, mock scanner trial (when available).
5. Noise-induced hearing loss or tinnitus.

   * Justification: individuals with noise-induced hearing problems may be particularly vulnerable to the acoustic noise generated by TMS and MRI equipment.
   * Screening tools: TMS safety screening.
6. Current use (any use in the past 4 weeks, chronic use within 6 past six months) of any investigational drug or of any medications with psychotropic, anti or pro-convulsive action.

   * Justification: The use of certain medications or drugs can lower seizure threshold and is therefore contraindicated for TMS.
   * Screening tools: MRI safety screening questionnaire and Medical history. A Urine toxicology that analyzes for presence of a broad range of prescription and nonprescription drugs may also be completed per the NIDA IRP screening protocol.
7. Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania.

   * Justification: The population of interest here is a healthy control population with no psychiatric disorders. In subjects with depression, bipolar disorder, mania or hypomania, there is a small chance that TMS can trigger (hypo)manic symptoms. Psychiatric symptoms could potentially alter BOLD signal.
   * Screening tools: structured psychiatric interview such as the MINI Screen Patient Questionnaire or Structured Clinical Interview for the DSM (SCID). Potential diagnoses will be further evaluated by a mental health professional.
8. Current use of nicotine or history more than about 20 cigarettes or 20 instances of nicotine use in lifetime or history of daily nicotine use.

   * Justification: The population of interest here is a healthy control population with no substance use disorder and therefore a minimal nicotine exposure history in the control group is required.
   * Screening tools: Self-report and CO < 6. A commercial urine cotinine test may also be used, with the expectation that results correspond to non-smoker status for the specific test being used, typically corresponding to a urine cotinine under about 20 ng/ml.
9. Meet current DSM-5 criteria for any substance use disorder, smoke daily, or urine toxicology positive for any illicit substance inconsistent with history given.

   * Justification: The population of interest here is a healthy control population with no substance use disorder. Current use of illicit substances could lower seizure threshold and is therefore contraindicated for TMS.
   * Screening tools: structured psychiatric interview such as the MINI Screen Patient Questionnaire or SCID (with SUD evaluation and potential follow up with a mental health professional), a drug use survey (DUS), and urine qualitative drug screen for common drugs of

   abuse. Participants who test positive at screening (under the NIDA IRP screening protocol) may be assessed for current intoxication. For participants who are not found to be currently intoxicated, screening staff will assess for SUD and coherence of their drug use history and toxicology with particular attention to substances for which they are positive and may require a return screening visit to demonstrate ability to produce a negative urine before allowing them to proceed to clearance for this study.
10. Have met DSM-5 criteria for any substance use disorder in the past.

    * Justification: the population of interest here is a healthy control population with no present or past substance use disorder.
    * Screening tools: structured psychiatric interview such as the MINI Screen Patient Questionnaire or SCID(with SUD evaluation and potential follow up evaluation with a mental health professional).
11. Pregnant individuals or those with reproductive potential who are sexually active and not using an acceptable form of contraception.

    * Justification: it is unknown whether TMS or MRI poses a risk to fetuses.
    * Screening tool: Medical assessments (urine pregnancy test) at the beginning of each visit that involves TMS or MRI.
12. Participation in an rTMS session less than two weeks ago.

    * Justification: in order to limit exposure to TMS, we will not enroll subjects who have received TMS less than two weeks ago.
    * Screening tool: TMS safety screening questionnaire.
13. History of learning disability, current ADHD or cognitive impairment

    * Justification: Cognitive impairment and learning disabilities are associated with alterations in brain regions and may introduce significant variably into the data.
    * Screening tool: self-report of special education classes, history of specific learning disability or mental retardation, and medical history. A validated IQ test such as Wechsler Abbreviated Scale of Intelligence (WASI) or Shipley-2 may also be completed.
14. Non-English Speaking

    * Justification: There is no direct benefit to participants in this study, and some of the study procedures involve more than minimal risk. To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify given the small sample size for each experiment. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI and TMS procedures. The inability to effectively communicate MRI and TMS safety procedures could compromise the safety of non-English speaking participants.
    * Screening tool: self-report.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
effects of TMS on fMRI blood oxygen level-dependent (BOLD) responses, TMS induced changes on resting state functional connectivity, and their associations with relevant structural connectivity revealed by DTI. | TMS visits
  fMRI blood oxygen level-dependent (BOLD) responses, TMS induced changes on resting state functional connectivity, and their associations with relevant structural connectivity revealed by DTI

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Yang, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Caparelli EC, Schleyer B, Zhai T, Gu H, Abulseoud OA, Yang Y. High-Frequency Transcranial Magnetic Stimulation Combined With Functional Magnetic Resonance Imaging Reveals Distinct Activation Patterns Associated With Different Dorsolateral Prefrontal Cortex Stimulation Sites. Neuromodulation. 2022 Jun;25(4):633-643. doi: 10.1016/j.neurom.2022.03.002. Epub 2022 Apr 10. PMID 35418339